CLINICAL TRIAL: NCT01496053
Title: Anti-inflammatory Effect of a Mushroom Extract (AndoSan)in Patients With Inflammatory Bowel Disease. A Prospective Study
Brief Title: Anti-inflammatory Effect of Agaricus Blazei Murill in Inflammatory Bowel Disease (IBD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: ImmunoPharma AS (Industry)
Responsible Party: Principal Investigator, Egil Johnson, MD, Phd, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AbM2012-IBD
Record Dates: First submitted 2011-12-15; First posted 2011-12-21 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Ulcerative Colitis; Crohn's Disease; Inflammatory Bowel Disease
Keywords: Cytokine levels in blood; Calprotectin in feces; Clinical symptom score.
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases | interventions — AndoSan; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AndoSan (Active Comparator): AndoSan given to IBD patients
  Interventions: Dietary Supplement: AndoSan
- Sugar extract (Sham Comparator): Sugar extract to IBD patients
  Interventions: Dietary Supplement: Sugar Extract

INTERVENTIONS:
Dietary Supplement: AndoSan — AndoSan 30 ml x 2 for 21 days
  Arms: AndoSan
Dietary Supplement: Sugar Extract — Sham comparator
  Arms: Sugar extract

SUMMARY:
Examine whether daily oral ingestion of a immunomodulatory mushroom extract (AndoSanTM) in patients with ulcerative colitis (UC) and Crohn's disease (CD), experience clinical, biochemical and genetical improvement in their disease.

A prospective randomised study comparing the mushroom extract with placebo.

ELIGIBILITY:
Inclusion Criteria:

* moderate disease

Exclusion Criteria:

* serious disease,
* biological treatment,
* pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Reduction in biochemical blood parameters (pro-inflammatory cytokines) | 21 days

SECONDARY OUTCOMES:
Reduction of calprotectin in feces. | 21 days
Clinical symptom score. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Egil Johnson, MD. Phd, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Oslo University Hospital, Ulleval, Oslo, Norway

REFERENCES:
- [Derived] Therkelsen SP, Hetland G, Lyberg T, Lygren I, Johnson E. Effect of the Medicinal Agaricus blazei Murill-Based Mushroom Extract, AndoSanTM, on Symptoms, Fatigue and Quality of Life in Patients with Crohn's Disease in a Randomized Single-Blinded Placebo Controlled Study. PLoS One. 2016 Jul 14;11(7):e0159288. doi: 10.1371/journal.pone.0159288. eCollection 2016. PMID 27415795
- [Derived] Therkelsen SP, Hetland G, Lyberg T, Lygren I, Johnson E. Effect of a Medicinal Agaricus blazei Murill-Based Mushroom Extract, AndoSan, on Symptoms, Fatigue and Quality of Life in Patients with Ulcerative Colitis in a Randomized Single-Blinded Placebo Controlled Study. PLoS One. 2016 Mar 2;11(3):e0150191. doi: 10.1371/journal.pone.0150191. eCollection 2016. PMID 26933886